CLINICAL TRIAL: NCT02182661
Title: A Phase III Long-term Study of Ba253BINEB in Patients With Bronchial Asthma
Brief Title: A Long-term Study of Ba253BINEB in Patients With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54.562
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- Ba253BINEB (Experimental)
  Interventions: Drug: Ba253BINEB

INTERVENTIONS:
Drug: Ba253BINEB

SUMMARY:
The objective of this study is to investigate the long-term safety of Ba253BINEB. Secondarily the long-term efficacy of Ba253BINEB is also investigated.

ELIGIBILITY:
Inclusion Criteria:

The patients with bronchial asthma and who satisfy the following criteria

1. Patients aged >= 20 years or older
2. Patients with mild to moderate severity
3. Patients must be able to understand the patient information form

Exclusion Criteria:

1. Patients who have taken an long acting corticosteroids(i.m.) within 1 month before the screening test
2. Patients using corticosteroid medication( p.o./ i.h.) at a dose in excess of the equivalent 10 mg/day of prednisolone
3. Patients with glaucoma
4. Patients who have prostatic hypertrophy
5. Patients with hypersensitivity to anticholinergic drugs
6. Patients who began treatment with hyposensitization or immunoregulator therapy within 3 month before the screening test
7. Patients complicated with chronic bronchitis, emphysema or bronchiectasis, making the assessment of drug efficacy against bronchial asthma difficult
8. Patients with serious hepatic disease, kidney disease or heart disorder and who are judged by the investigator as inappropriate as the subjects of study
9. Women who are pregnant or who may become pregnant, or nursing women
10. Patients who are judged by the investigator as inappropriate as the subjects of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 1998-07; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 30 weeks
Number of patients with abnormal changes in blood pressure and heart rate | Baseline, up to 28 weeks
Number of patients with abnormal changes in ECG (electrocardiogram) | Baseline, up to 28 weeks
Number of patients with abnormal changes in laboratory parameters | Baseline, up to 28 weeks

SECONDARY OUTCOMES:
Change from baseline in symptom score | Baseline, up to 28 weeks
Change from baseline in treatment score | Baseline, up to 28 weeks
Change from baseline in asthma score | Baseline, week 28
Change from baseline in daily life score | Baseline, up to 28 weeks
Change from baseline in nocturnal sleep score | Baseline, up to 28 weeks
Change from baseline in Peak expiratory flow rate (PEFR) | Baseline, up to 28 weeks
Physician's global evaluation (overall improvement and final overall improvement) | Baseline, up to 28 weeks
Patient's impression | Week 28
Change from baseline in FEV1 (Forced expiratory volume in one second) | Baseline, up to 28 weeks
Change from baseline in FVC (Forced vital capacity) | Baseline, up to 28 weeks